CLINICAL TRIAL: NCT00132015
Title: A Phase II Clinical Trial of 17-(Allylamino)-17- Demethoxygeldanamycin (17-AAG, NSC 330507 and EPL Diluent, NSC 704057) in Adults With Systemic Mastocytosis
Brief Title: 17-N-Allylamino-17-Demethoxygeldanamycin in Treating Patients With Systemic Mastocytosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institutes of Health Clinical Center (CC) (NIH)
Collaborators: National Cancer Institute (NCI) (NIH)
Masking: None | Purpose: Treatment
Other Study IDs: 060076; 06-C-0076; NCI-6454; NCI-P6175; CDR0000438778; NCT00285311 (obsolete NCT alias)
Record Dates: First submitted 2005-08-16; First posted 2005-08-19 (Estimated); Last update posted 2012-03-15 (Estimated); Status verified 2012-03

CONDITIONS: Chronic Myeloproliferative Disorders; Leukemia; Lymphoma; Nonneoplastic Condition; Precancerous Condition
Keywords: Waldenström macroglobulinemia; multicentric Castleman disease; unicentric Castleman disease; adult grade III lymphomatoid granulomatosis; polycythemia vera; essential thrombocythemia; hairy cell leukemia; monoclonal gammopathy of undetermined significance; adult Burkitt lymphoma; adult diffuse large cell lymphoma; adult diffuse mixed cell lymphoma; adult diffuse small cleaved cell lymphoma; adult immunoblastic large cell lymphoma; adult lymphoblastic lymphoma; grade 1 follicular lymphoma; grade 2 follicular lymphoma; grade 3 follicular lymphoma; mantle cell lymphoma; marginal zone lymphoma; small lymphocytic lymphoma; precancerous condition
MeSH Terms: conditions — Myeloproliferative Disorders; Leukemia; Lymphoma; Precancerous Conditions; Waldenstrom Macroglobulinemia; Multi-centric Castleman's Disease; Angiolymphoid Hyperplasia with Eosinophilia; Polycythemia Vera; Thrombocythemia, Essential; Leukemia, Hairy Cell; Monoclonal Gammopathy of Undetermined Significance; Burkitt Lymphoma; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Non-Hodgkin; Lymphoma, Large-Cell, Immunoblastic; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma, Follicular; Lymphoma, Mantle-Cell; Lymphoma, B-Cell, Marginal Zone; Leukemia, Lymphocytic, Chronic, B-Cell | interventions — tanespimycin

INTERVENTIONS:
Drug: tanespimycin

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as 17-N-allylamino-17-demethoxygeldanamycin (17-AAG), work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing.

PURPOSE: This phase II trial is studying how well 17-AAG works in treating patients with systemic mastocytosis.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the efficacy of 17-N-allylamino-17-demethoxygeldanamycin (17-AAG), in terms of decreases in the number of mast cells in the bone marrow and in serum tryptase levels, in patients with systemic mastocytosis.

Secondary

* Determine the quality of life of patients treated with this drug.
* Determine hematological and non-hematological toxicity of this drug in these patients.

OUTLINE: This is a multicenter study.

Patients receive 17-N-allylamino-17-demethoxygeldanamycin (17-AAG) IV over 2-6 hours on days 1, 4, 8, and 11. Treatment repeats every 21 days for at least 6 courses in the absence of disease progression or unacceptable toxicity. Patients achieving a complete response (CR) receive at least 2 additional courses beyond CR. Patients achieving a partial response receive at least 4 additional courses beyond their maximum response. Selected patients may receive additional courses of therapy beyond the protocol guidelines at the discretion of the principal investigator.

Quality of life is assessed at baseline and before each treatment course.

PROJECTED ACCRUAL: A total of 12-37 patients will be accrued for this study within approximately 10-18 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed systemic mastocytosis

  * Objective evidence of disease, as defined by the following:

    * Hemoglobin < 10 g/dL
    * Recurrent mast cell mediator-release symptoms that impair the patient's quality of life
    * Symptomatic hepatosplenomegaly
    * Ascites
    * Symptomatic bone disease
    * Profound constitutional symptoms (e.g., fatigue, asthenia, flushing, hyperpyrexia, weight loss, myalgia, and arthralgia)
    * Elevated serum tryptase level
* Mast cell leukemia allowed
* Mastocytosis associated with myeloproliferative disease (e.g., hypereosinophilic syndrome or chronic myelomonocytic leukemia) allowed
* Patients with eosinophilia (i.e., absolute eosinophil count ≥ 1,000/mm^3) must be evaluated for the presence or absence of FIP1L1-PDGFRA mutation; if the mutation is absent, the patient is eligible; if the mutation is present, the patient is eligible provided disease is refractory to imatinib mesylate
* Patients with indolent disease must have a serum tryptase level ≥ 50 ng/mL OR episodes of anaphylaxis that occur with a frequency of > 1 per month

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* ECOG 0-2

Life expectancy

* At least 3 months

Hematopoietic

* See Disease Characteristics
* Platelet count ≥ 100,000/mm^3 (> 25,000/mm^3 for patients with organomegaly)
* Absolute granulocyte count ≥ 1,500/mm^3(> 750/mm^3 for patients with organomegaly)

Hepatic

* AST and ALT ≤ 2 times upper limit of normal (ULN) (< 4 times ULN for patients with hepatomegaly)
* Bilirubin normal
* Alkaline phosphatase ≤ 3 times ULN

Renal

* Creatinine ≤ 1.4 mg/dL OR
* Creatinine clearance ≥ 60 mL/min

Cardiovascular

* No New York Heart Association class III-IV congestive heart failure
* No history of myocardial infarction within the past year
* No history of uncontrolled dysrhythmia
* No uncontrolled angina
* No ischemic heart disease within the past 12 months
* No congenital long QT syndrome
* No left bundle branch block
* No serious ventricular arrhythmia (ventricular tachycardia or ventricular fibrillation ≥ 3 beats in a row)
* QTc interval < 450 msec for males or 470 msec for females
* LVEF > 40% by MUGA
* MUGA or echocardiogram normal
* No prior history of cardiac toxicity after receiving anthracyclines (e.g., doxorubicin hydrochloride, daunorubicin hydrochloride, mitoxantrone hydrochloride, bleomycin, or carmustine)
* No cardiac symptoms ≥ grade 2
* No other significant cardiac disease

Pulmonary

* No symptomatic pulmonary disease requiring medication including any of the following:

  * Dyspnea on or off exertion
  * Paroxysmal nocturnal dyspnea
  * Requirement for oxygen
  * Significant pulmonary disease (e.g., chronic obstructive/restrictive pulmonary disease)
* No home oxygen meeting the Medicare requirement
* No compromised pulmonary status (i.e., DLCO ≤ 80%)
* No prior history of pulmonary toxicity after receiving anthracyclines (e.g., doxorubicin hydrochloride, daunorubicin hydrochloride, mitoxantrone hydrochloride, bleomycin, or carmustine)
* No pulmonary symptoms ≥ grade 2

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for ≥ 6 months after completion of study treatment
* HIV negative
* No active uncontrolled infection
* No serious medical illness
* No other non-malignant systemic disease
* No history of serious allergic reaction to eggs
* No other malignancy within the past 2 years except dermatological cancer

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* At least 4 weeks since prior chemotherapy

Endocrine therapy

* Steroids allowed provided tapering to the lowest level possible to treat thrombocytopenia, diarrhea, or malabsorption symptoms of systemic mastocytosis

Radiotherapy

* At least 4 weeks since prior radiotherapy
* No prior radiation that included the heart in the field (e.g., mantle) or chest

Surgery

* Not specified

Other

* At least 4 weeks since prior tyrosine kinase inhibitors
* No concurrent complimentary or alternative medications* including, but not limited to, the following:

  * Hypericum perforatum (St. John's wort)
  * Milk thistle
  * Kava kava
  * Mistletoe extract
* No concurrent agents that cause QTc prolongation
* No concurrent antiarrhythmic therapy
* No other concurrent investigational therapy NOTE: *Unless approved by the investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Estimated)
Dates: Start 2006-05; Primary Completion 2007-12 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
Objective response (complete and partial response)

SECONDARY OUTCOMES:
Quality of life as assessed by the European Organization for Research of the Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ-C30) at baseline and prior to each treatment course

CONTACTS AND LOCATIONS:
Overall Officials: Antonio T. Fojo, MD, PhD, Principal Investigator — National Cancer Institute (NCI)
Locations (2):
- United States (2):
  - Warren Grant Magnuson Clinical Center - NCI Clinical Trials Referral Office, Bethesda, Maryland
  - NCI - Center for Cancer Research, Bethesda, Maryland